CLINICAL TRIAL: NCT01928264
Title: Physical Activity in Insurance Medicine: Effects on Psycho(-Physio-)Logical Functions, Capacity / Participation Skills, and the Ability to Work in Psychiatric Disorders
Brief Title: Physical Activity in Insurance Medicine: Effects on Patients With Psychiatric Disorders
Acronym: PhysActIV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Psychiatric Hospital of the University of Basel (Other); Institute for Exercise and Health Sciences, University of Basle, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114/13
Record Dates: First submitted 2013-08-05; First posted 2013-08-23 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Depressive Disorder; Somatoform Disorder; Anxiety Disorder; Personality Disorder
Keywords: Mental disorders; Physical activity; Disability pension; Disability pension due to mental illness; Ability to work; Mental toughness
MeSH Terms: conditions — Depressive Disorder; Somatoform Disorders; Anxiety Disorders; Personality Disorders; Mental Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity (Experimental): Physical activity group program over 12 weeks; 1 hour sessions, 2 times a week
  Interventions: Behavioral: Physical activity
- Leisure time activities (No Intervention): Predominantly sedentary leisure time group activities, like playing board games, doing handicrafts, etc.; 12 weeks, 1 hour sessions, 2 times a week

INTERVENTIONS:
Behavioral: Physical activity
  Arms: Physical activity

SUMMARY:
We will conduct a randomized control trial to investigate whether and to what extent regular and guided group physical activity over 12 weeks (2 sessions à 1 hour/week) improves physical fitness and (physio-)psychological functions (like subjective sleep, mental toughness, perceived stress, self-efficacy, etc.), as well as participation skills and the ability to work, in claimants for a disability pension due to psychiatric disorders, whose ability to work had recently been assessed by means of a psychiatric expert opinion. The control group is designed very similar and implies predominantly sedentary leisure time group activities (e.g. playing board games, doing handicrafts). Measures will be performed at baseline, post-test, and at follow ups three and twelve months after post-test, some variables will additionally be assessed 4-weekly during the intervention. We expect that intervention group participants will report and show, respectively, more improved physical fitness, (physio-)psychological functioning and participations skills, as well as increased ability to work, compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Claimants for a disability pension due to a mental disorder, whose ability to work has been recently assessed by means of a psychiatric expert opinion
* Both genders
* 18-55 years old
* Clinical diagnosis of depressive disorder, somatoform disorder, anxiety disorder, personality disorder
* Sufficient competence in understanding, speaking and reading German
* Sufficient cognitive, emotional and social level of functioning to be able to participate in a group
* Physical Activity Readiness Questionnaire without evidence for reduction
* or: Physical activity readiness certificated by the general practitioner
* Informed consent

Exclusion Criteria:

* Comorbidity with a somatic disorder that limits the ability for physical exercises
* Pregnancy
* Ongoing disturbance of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in the ability to work (h/d / %) | baseline and 15 months

SECONDARY OUTCOMES:
Change in the ability to work (h/d / %) | baseline and 6 months
Change in the ability to work (h/d / %) | baseline and 12 weeks
Change in participation skills (sum score) | baseline and 15 months
Change in participation skills (sum score) | baseline and 6 months
Change in participation skills (sum score) | baseline and 12 weeks
Change in psychological functioning (sum scores) | baseline and 15 months
Change in psychological functioning (sum scores) | baseline and 6 months
Change in psychological functioning (sum scores) | baseline and 12 weeks
Change in subjective sleep quality (sum score) | baseline and 15 months
Change in subjective sleep quality (sum score) | baseline and 6 months
Change in subjective sleep quality (sum score) | baseline and 12 weeks
Change in subjective sleep quality (sum score) | baseline and 8 weeks
Change in subjective sleep quality (sum score) | baseline and 4 weeks
Change in subjectively perceived stress (sum score) | baseline and 15 months
Change in subjectively perceived stress (sum score) | baseline and 6 months
Change in subjectively perceived stress (sum score) | baseline and 12 weeks
Change in subjectively perceived stress (sum score) | baseline and 8 weeks
Change in subjectively perceived stress (sum score) | baseline and 4 weeks
Change in Clinical Global Impression (sum score) | baseline and 15 months
Change in Clinical Global Impression (sum score) | baseline and 6 months
Change in Clinical Global Impression (sum score) | baseline and 12 weeks
Change in Leisure-time physical activity (sum score) | baseline and 15 months
Change in Leisure-time physical activity (sum score) | baseline and 6 months
Change in Leisure-time physical activity (sum score) | baseline and 12 weeks
Change in self-efficacy (sum score) | baseline and 15 months
Change in self-efficacy (sum score) | baseline and 6 months
Change in self-efficacy (sum score) | baseline and 12 weeks
Change in self-efficacy (sum score) | baseline and 8 weeks
Change in self-efficacy (sum score) | baseline and 4 weeks

OTHER OUTCOMES:
Change in physical fitness (VO2max = ml/kg/min) | baseline and 15 months
Change in physical fitness (VO2max = ml/kg/min) | baseline and 6 months
Change in physical fitness (VO2max = ml/kg/min) | baseline and 12 weeks
Change in physical fitness (VO2max = ml/kg/min) | baseline and 8 weeks
Change in physical fitness (VO2max = ml/kg/min) | baseline and 4 weeks
Change in perceived fitness (sum score) | baseline and 15 months
Change in perceived fitness (sum score) | baseline and 6 months
Change in perceived fitness (sum score) | baseline and 12 weeks
Change in perceived fitness (sum score) | baseline and 8 weeks
Change in perceived fitness (sum score) | baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Rabovsky, MD, Principal Investigator — Psychiatric Hospital of the University of Basel
Locations (1):
- Psychiatric Hospital of the University of Basel, Basel, Switzerland